CLINICAL TRIAL: NCT01198392
Title: A Clinical Trial of S-1 Plus Cisplatin Versus 5-FU Plus Cisplatin in Patients With Unresectable or Advanced Gastric Cancer
Brief Title: Trial of S-1 Plus Cisplatin in Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Zhongzhen Guan ,Ruihua Xu, Sun Yat-sen University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005L02859
Record Dates: First submitted 2010-09-01; First posted 2010-09-10 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2008-08

CONDITIONS: Gastric Cancer
Keywords: gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S-1 plus cisplatin; Tegafur; gimeracil; potassium oxonate; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-1 plus cisplatin (Experimental): S-1:80 mg/m2/day po twice daily on Day 1-21,cisplatin: 20mg/m2 iv on Day 1-4, repeat every 5 weeks.Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: s-1 plus cisplatin
- 5-Fu plus cisplatin (Active Comparator): 5-Fu 800 mg/m2/d CI 120h ,Cisplatin 20 mg/m2 as a 2 hour i.v. infusion(on day 1 to day 4 )repeat every 4 weeks.Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: 5-Fu plus cisplatin

INTERVENTIONS:
Drug: s-1 plus cisplatin — S-1:80 mg/m2/day po twice daily on Day 1-21,cisplatin: 20mg/m2 iv on Day 1-4, repeat every 5 weeks. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Tegafur,Gimeracil and Oteracil Potassium Capsules
  Arms: S-1 plus cisplatin
Drug: 5-Fu plus cisplatin — 5-Fu 800 mg/m2/d CI 120h ,Cisplatin 20 mg/m2 as a 2 hour i.v. infusion(on day 1 to day 4 )repeat every 4 weeks.
  Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: 5-fluoroura
  Arms: 5-Fu plus cisplatin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of s-1 plus cisplatin versus 5-FU plus cisplatin as first-line therapy in the treatment of patients with advanced gastric cancer.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label,multicenter study. Patients are randomized to one of two treatment arms : S-1 plus cisplatin and 5-FU plus cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach with inoperable locally advanced or recurrent and/or metastatic disease.
* Male or female.
* Age 18 -75.
* Previous chemotherapy for advanced/metastatic disease (prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study).
* Measurable disease, according to the Response Evaluation Criteria in Solid Tumours(RECIST)
* ECOG Performance status 0, 1 or 2
* Haematological, Biochemical and Organ Function: Neutrophil count >2.0 × 10 9/L, platelet count > 100 ×10 9/L. Serum bilirubin< 1.5 × upper limit of normal (ULN); or, AST or ALT < 2.5 × ULN (or < 5 × ULN in patients with liver metastases); or, alkaline phosphatase< 2.5 × ULN (or > 5 × ULN in patients with liver metastases,Creatinine clearance > 60 mL/min.
* Signed informed consent.

Exclusion Criteria:

* prior adjuvant/neoadjuvant therapy more than two regiments.
* Received any investigational drug treatment within 30 days of start of study treatment.
* Patients with active gastrointestinal bleeding.
* Neurological toxicity ≥ grade 2 NCI-CTCAE.
* Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma.
* History or clinical evidence of brain metastases.
* Serious uncontrolled systemic intercurrent illness, e.g. infections or poorly controlled diabetes.
* Pregnancy women.
* Subjects with reproductive potential not willing to use an effective method of contraception.
* Patients with known active infection with HIV.
* Known hypersensitivity to any of the study drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression | The time from randomization until objective tumor progression or death

SECONDARY OUTCOMES:
Response rate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: RUIHUA XU, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Gangdong, China

REFERENCES:
- [Derived] Li YH, Qiu MZ, Xu JM, Sun GP, Lu HS, Liu YP, Zhong MZ, Zhang HL, Yu SY, Li W, Hu XH, Wang JJ, Cheng Y, Zhou JT, Guo ZQ, Guan ZG, Xu RH. S-1 plus cisplatin versus fluorouracil plus cisplatin in advanced gastric or gastro-esophageal junction adenocarcinoma patients: a pilot study. Oncotarget. 2015 Oct 27;6(33):35107-15. doi: 10.18632/oncotarget.5959. PMID 26439700